CLINICAL TRIAL: NCT04357925
Title: Quality of Life in Prostate Cancer Patients: Challenges and Prospects for Reducing Disparities in the Caribbean
Brief Title: Quality of Life in Prostate Cancer Patients
Acronym: QoLProstateMQ
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 19_RIPH3_08; 2019-A02116-51 (Other: ANSM)
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Public Health; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recording cancer data in cancer registries is essential for producing reliable population-based data for service planning, monitoring and evaluation. Prostate cancer (PCa) remains the most frequent type of cancer in terms of incidence and mortality in men in the Caribbean. The quality of life PCa cohort will assess quality of life and patient outcomes in Martinique using a digital platform for patient-reported outcome measures.

DETAILED DESCRIPTION:
The Martinique Cancer Registry database is the largest clinical database among the French population-based cancer registries in the Caribbean, including more than 38 000 cancer cases, with 1650 new cancer cases per year, including 550 new PCa cases per year (2010-2014 latest period). In 2020, follow-up will include vital status, assessment of quality of life with the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) Core 30 and the Prostate cancer module QLQ-PR25. Urinary incontinence and erectile dysfunction recorded prior to treatment will be analysed 1, 3 and 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years and residing in Martinique, with prostate cancer diagnosed from 2020
* The patient has provided informed consent
* Patient with social security coverage

Exclusion Criteria:

* Refusal to participate
* Patient with a second cancer, five years after diagnosis
* Patient who could not answer the quality of life questionnaires
* Patient not fluent in French
* Person under legal protection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer diagnosed in Martinique in differents units care.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of overall Quality of Life: Questionnaire | At the date of diagnosis of the disease, at 1 year, 3 years and 5 years
  Change of quality of life questionnaire related to sexual dysfunction
Evaluation of overall Quality of Life: Questionnaire | At the date of diagnosis of the disease, at 1 year, 3 years and 5 years
  Change of quality of life questionnaire related to urinary troubles

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse CONTARET-JOACHIM, Study Director — CHU Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique